CLINICAL TRIAL: NCT05595252
Title: Retrospective Study on the Evolution of CIN 1 to 3 in Per and Postpartum in Nancy From 2014 to 2022
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, MARTIN Elena, Assistant clinical Director, Central Hospital, Nancy, France
Other Study IDs: 2022PI157/EUDRACT
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CIN lésions during pregnancy
  Interventions: Biological: cervical biopsy

INTERVENTIONS:
Biological: cervical biopsy — cervical biopsy made during and after pregancy

SUMMARY:
In France, the screening rate for cervical cancer remains too low. Screening is simple and non-invasive.

Pregnant patients are most of the time young and are part of the target population for screening, and for many women, it is the first encounter with a gynecologist.

The cervical smear is therefore an important step of the first consultation during pregnancy In the case of pathological results, colposcopies with biopsies are performed, frequently finding CIN 1 to 3. (cervical intraepithelial neoplasia) These CIN lesions evolve slowly and most of the time, treatment can be withheld until the end of the pregnancy.

Several studies suggest a higher regression rate in pregnant patients. Our study will evaluate the rate of regression, progression or persistence of these lesions in per and post partum patients in Nancy, between 2014 and 2022.

To obtain our results, we will compare the results of per and post partum biopsies in each patient.

In a second step, we will study the risk factors of aggravation or on the contrary the protective factors, allowing a faster regression of the lesions

ELIGIBILITY:
Inclusion Criteria:

* women who have a CIN lesion during pregnancy
* in Nancy, France, MRUN Center
* between 2014 and 2022

Exclusion Criteria:

* lost of follow up women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: study on patients who were pregnant and have a CIN lesion at the same time, care at the MRUN, the Nancy Régional Maternity between 2014 and 2022
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
progress, persistence or regression of CIN lesion count | up to one year after delivery
  cervical biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Camille BENOIT, Principal Investigator — CHRU Nancy
Locations (1):
- BENOIT Camille, Nancy, France